CLINICAL TRIAL: NCT00221013
Title: Multicentre, Unblinded, Open Label, Randomised, Controlled Trial to Assess the Effect of Augmented Vs. Normal Continuous Renal Replacement Therapy (CRRT) on 90-Day All-Cause Mortality of Intensive Care Unit Patients With Severe Acute Renal Failure (ARF).
Brief Title: Augmented Vs. Normal Renal Replacement Therapy in Severe Acute Renal Failure (ARF).
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The George Institute (Other)
Collaborators: ANZICS Clinical Trials Group (Network)
Responsible Party: Project Manager, The George Institute
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: GI-RE-ARF001-40-R; 352550
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2009-02-27 (Estimated); Status verified 2009-02

CONDITIONS: Acute Renal Failure
Keywords: Acute Renal Failure; Continuous Renal Replacement Therapy; Continuous Veno-Venous Haemofiltration; Continuous Veno-Venous Haemodiafiltration; Renal Replacement Therapy
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Higher intensity CRRT regimen (Experimental)
  Interventions: Procedure: "augmented" CRRT regimen
- Lower intensity CRRT regimen (Active Comparator)
  Interventions: Procedure: "augmented" CRRT regimen

INTERVENTIONS:
Procedure: "augmented" CRRT regimen — We randomly assigned critically ill patients with acute kidney injury to receive CRRT in the form of post-dilution continuous veno-venous hemodiafiltration (CVVHDF) at 25 ml/kg/hr (lower intensity) or 40 ml/kg/hr (higher intensity) of effluent flow.

SUMMARY:
This study seeks to determine if increasing the dose of continuous renal replacement therapy (CRRT) reduces 90-day all cause mortality in Intensive Care Unit (ICU) patients with severe acute renal failure (ARF).

DETAILED DESCRIPTION:
Study Title - Multicentre, Unblinded, Randomised, Controlled Trial to assess the effect of Augmented vs. Normal Continuous Renal Replacement Therapy (CRRT) on 90-day all-cause mortality of Intensive Care Unit Patients with Severe Acute Renal Failure (ARF).

Clinical Phase - IV

Study Rationale - This study will provide high quality evidence from a mulit-center randomised controlled trial about the comparative effects of different targets for CRRT dose in patients with ARF treated in the Australasian intensive care setting. This evidence will have direct relevance to decisions about the care of critically ill patients admitted to intensive care units in Australia and New Zealand. If this study confirms the treatment effect reported in the Lancet study, augmented dose CRRT is likely too become the standard of treatment, saving 250-300 lives/year in Australia and 15,000 lives/year worldwide.

Trial Design - The proposed study will compare an "augmented" CRRT regimen to deliver an effluent rate of 40 ml/kg/hr compared to "normal" CRRT at an effluent rate of 25ml/kg/hr in ICU patients with severe ARF.

Subject Participation - 90 days

Rationale for Number of Subjects - Assuming a 90-day mortality rate of 60% in our control group the study of 1,500 patients will have 90% power of detecting an 8.5% absolute reduction from a 90-day mortality of 60% in the control group to 51.5% in the intervention group (P<0.05).

Approximate duration of Study - 36 months

Study Objective(s)

Primary - The primary study outcome is death from all causes at 90 days after randomisation.

Secondary

* Death within the in the intensive care unit.
* Death within 28 days of randomisation.
* Death prior to hospital discharge.
* Length of ICU stay.
* Length of hospital stay.
* The need for and duration of other organ support (inotropic/vasopressor support and positive pressure ventilation).
* CRRT-free days.
* Dialysis-independent survival.

Criteria for Inclusion

1. The treating clinician believes that the patient requires CRRT for acute renal failure.
2. The clinician is uncertain about the balance of benefits and risks likely to be conferred by treatment with higher intensity or lower intensity CRRT.
3. The treating clinicians anticipate treating the patient with CRRT for at least 72 hours.
4. Informed consent has been obtained
5. The patient fulfils at least ONE of the following clinical criteria for initiating CRRT:

   1. Oliguria (urine output < 100ml/6hr) that has been unresponsive to fluid resuscitation measures.
   2. Hyperkalemia ([K+] > 6.5 mmol/L).
   3. Severe acidemia (pH < 7.2).
   4. Urea > 25 mmol/liter.
   5. Creatinine >300 micromol/L in the setting of ARF.
   6. Clinically significant organ oedema in the setting of ARF (eg: lung).

Criteria for Exclusion

1. Patient age is <18 years.
2. Death is imminent (<24 hours).
3. There is a strong likelihood that the study treatment would not be continued in accordance with the study protocol.
4. The patient has been treated with CRRT or other dialysis previously during the same hospital admission.
5. The patient was on maintenance dialysis prior to the current hospitalisation.
6. The patient's body weight is <60 kg or >120kg.
7. Any other major illness that, in the investigator's judgment, will substantially increase the risk associated with the subject's participation in this study.

Approximate Number of Subjects - 1500

Approximate Number of Study Centres - 35 centres distributed in both Australia and New Zealand will participate in the study.

Treatment Administration - Each participant will be randomised to receive CRRT in the technical form of CVVHDF either at an intensity of 25ml/kg/hr of effluent flow(normal CRRT) or 40 ml/kg/hr of effluent flow (augmented CRRT).

Safety Evaluation - Safety for individual patients will be assessed on an ongoing basis by physical examination, including vital signs, outputs from dialysis machine records, laboratory assessments, and monitoring of adverse events. Overall study safety will be ensured by an Independent Data Safety Monitoring Committee, independent from all Trial investigators, which will perform ongoing review of predefined safety parameters and study conduct.

Efficacy Evaluation - Overall survival at 90 days post randomisation

Statistical Analysis - The interim analyses will be conducted when approximately 500 and 1000 patients have completed 90 day follow up, as dictated by the Data Safety Monitoring Committee. The final analysis will occur when outcome data for the target 1500 subjects is available. At interim and final analysis, the baseline and outcome variables will be compared using Students t test, Chi squared and the Mann-Whitney U test as appropriate. Survival analysis will be assessed using the Mantel-Cox test. The final statistical analysis will be performed according to a pre-determined statistical analysis plan (Critical Care and Resuscitation, 2009 in press).

ELIGIBILITY:
Inclusion Criteria:

1. The treating clinician believes that the patient requires CRRT for acute renal failure.
2. The clinician is uncertain about the balance of benefits and risks likely to be conferred by treatment with higher intensity or lower intensity CRRT.
3. The treating clinicians anticipate treating the patient with CRRT for at least 72 hours.
4. Informed consent has been obtained
5. The patient fulfils ONE of the following clinical criteria for initiating CRRT:

   * Oliguria (urine output < 100ml/6hr) that has been unresponsive to fluid resuscitation measures.
   * Hyperkalemia ([K+] > 6.5 mmol/L).
   * Severe acidemia (pH < 7.2).
   * Urea > 25 mmol/liter.
   * Creatinine >300 micromol/L in the setting of ARF.
   * Clinically significant organ oedema in the setting of ARF (eg: lung).

Exclusion Criteria:

1. Patient age is <18 years.
2. Death is imminent (<24 hours).
3. There is a strong likelihood that the study treatment would not be continued in accordance with the study protocol.
4. The patient has been treated with CRRT or other dialysis previously during the same hospital admission.
5. The patient was on maintenance dialysis prior to the current hospitalisation.
6. The patient's body weight is <60 kg or >100kg.
7. Any other major illness that, in the investigator's judgment, will substantially increase the risk associated with the subject's participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1508 (Actual)
Dates: Start 2005-11; Primary Completion 2008-10 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Death from all causes at 90 days after randomisation. | Within 90 days after randomisation

SECONDARY OUTCOMES:
Death within the in the intensive care unit. | 0 to 90 days
Death within 28 days of randomisation. | Within 28 days of randomisation.
Death prior to hospital discharge. | 0 to 90 days
Length of ICU stay. | 0 to 90 days
Length of hospital stay. | 0 to 90 days
The need for and duration of other organ support (inotropic/vasopressor support and positive pressure ventilation). | 0 to 90 days
CRRT-free days. | 0 to 90 days
Dialysis-independent survival. | 0 to 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Prof Rinaldo Bellomo, MD, Study Chair — Austin Hospital, Melbourne Australia; Alan Cass, MD, Principal Investigator — The George Institute; Simon Finfer, MD, Principal Investigator — Royal North Shore Hospital; Carlos Scheinkestel, MD, Principal Investigator — The Alfred; Robyn Norton, MD, Principal Investigator — The George Institute; John Myburgh, MD, Principal Investigator — St George Hospital (Sydney); Louise Cole, MD, Principal Investigator — Nepean Blue Mountains Local Health District; Martin Gallagher, MD, Principal Investigator — The George Institute; Shay McGuinness, MD, Principal Investigator — Auckland City Hospital CVICU; Colin McArthur, MD, Principal Investigator — Auckland City Hospital DCCM
Locations (1):
- The Austin Hopsital, Heidelberg, Victoria, Australia

REFERENCES:
- [Background] RENAL Study Investigators. Renal replacement therapy for acute kidney injury in Australian and New Zealand intensive care units: a practice survey. Crit Care Resusc. 2008 Sep;10(3):225-30. PMID 18798721
- [Background] RENAL Study Investigators; Bellomo R, Cass A, Cole L, Finfer S, Gallagher M, Goldsmith D, Myburgh J, Norton R, Scheinkestel C. Design and challenges of the Randomized Evaluation of Normal versus Augmented Level Replacement Therapy (RENAL) Trial: high-dose versus standard-dose hemofiltration in acute renal failure. Blood Purif. 2008;26(5):407-16. doi: 10.1159/000148400. PMID 18856012
- [Derived] Fayad AI, Buamscha DG, Ciapponi A. Timing of kidney replacement therapy initiation for acute kidney injury. Cochrane Database Syst Rev. 2022 Nov 23;11(11):CD010612. doi: 10.1002/14651858.CD010612.pub3. PMID 36416787
- [Derived] Naorungroj T, Neto AS, Wang A, Gallagher M, Bellomo R. Renal outcomes according to renal replacement therapy modality and treatment protocol in the ATN and RENAL trials. Crit Care. 2022 Sep 6;26(1):269. doi: 10.1186/s13054-022-04151-5. PMID 36068554
- [Derived] Tsujimoto Y, Miki S, Shimada H, Tsujimoto H, Yasuda H, Kataoka Y, Fujii T. Non-pharmacological interventions for preventing clotting of extracorporeal circuits during continuous renal replacement therapy. Cochrane Database Syst Rev. 2021 Sep 14;9(9):CD013330. doi: 10.1002/14651858.CD013330.pub2. PMID 34519356
- [Derived] Serpa Neto A, Naorungroj T, Murugan R, Kellum JA, Gallagher M, Bellomo R. Heterogeneity of Effect of Net Ultrafiltration Rate among Critically Ill Adults Receiving Continuous Renal Replacement Therapy. Blood Purif. 2021;50(3):336-346. doi: 10.1159/000510556. Epub 2020 Oct 7. PMID 33027799
- [Derived] Murugan R, Kerti SJ, Chang CH, Gallagher M, Clermont G, Palevsky PM, Kellum JA, Bellomo R. Association of Net Ultrafiltration Rate With Mortality Among Critically Ill Adults With Acute Kidney Injury Receiving Continuous Venovenous Hemodiafiltration: A Secondary Analysis of the Randomized Evaluation of Normal vs Augmented Level (RENAL) of Renal Replacement Therapy Trial. JAMA Netw Open. 2019 Jun 5;2(6):e195418. doi: 10.1001/jamanetworkopen.2019.5418. PMID 31173127
- [Derived] Wang AY, Trongtrakul K, Bellomo R, Li Q, Cass A, Gallagher M; RENAL Study Investigators and the ANZICS Clinical Trials Group. HMG-CoA reductase inhibitors (statins) and acute kidney injury: A secondary analysis of renal study outcomes. Nephrology (Carlton). 2019 Sep;24(9):912-918. doi: 10.1111/nep.13597. Epub 2019 May 27. PMID 31058387
- [Derived] Roberts DM, Liu X, Roberts JA, Nair P, Cole L, Roberts MS, Lipman J, Bellomo R; RENAL Replacement Therapy Study Investigators. A multicenter study on the effect of continuous hemodiafiltration intensity on antibiotic pharmacokinetics. Crit Care. 2015 Mar 13;19(1):84. doi: 10.1186/s13054-015-0818-8. PMID 25881576
- [Derived] Wang AY, Bellomo R, Ninomiya T, Lo S, Cass A, Jardine M, Gallagher M; RENAL Study Investigators; ANZICS Clinical Trials Group. Angiotensin-converting enzyme inhibitor usage and acute kidney injury: a secondary analysis of RENAL study outcomes. Nephrology (Carlton). 2014 Oct;19(10):617-22. doi: 10.1111/nep.12284. PMID 24894685
- [Derived] Bellomo R, Cass A, Cole L, Finfer S, Gallagher M, Lee J, Lo S, McArthur C, McGuinness S, Myburgh J, Norton R, Scheinkestel C; RENAL Study Investigators; Su S. Calorie intake and patient outcomes in severe acute kidney injury: findings from The Randomized Evaluation of Normal vs. Augmented Level of Replacement Therapy (RENAL) study trial. Crit Care. 2014 Mar 14;18(2):R45. doi: 10.1186/cc13767. PMID 24629036
- [Derived] Gallagher M, Cass A, Bellomo R, Finfer S, Gattas D, Lee J, Lo S, McGuinness S, Myburgh J, Parke R, Rajbhandari D; POST-RENAL Study Investigators and the ANZICS Clinical Trials Group. Long-term survival and dialysis dependency following acute kidney injury in intensive care: extended follow-up of a randomized controlled trial. PLoS Med. 2014 Feb 11;11(2):e1001601. doi: 10.1371/journal.pmed.1001601. eCollection 2014 Feb. PMID 24523666
- [Derived] Bellomo R, Lipcsey M, Calzavacca P, Haase M, Haase-Fielitz A, Licari E, Tee A, Cole L, Cass A, Finfer S, Gallagher M, Lee J, Lo S, McArthur C, McGuinness S, Myburgh J, Scheinkestel C; RENAL Study Investigators and ANZICS Clinical Trials Group. Early acid-base and blood pressure effects of continuous renal replacement therapy intensity in patients with metabolic acidosis. Intensive Care Med. 2013 Mar;39(3):429-36. doi: 10.1007/s00134-012-2800-0. Epub 2013 Jan 11. PMID 23306586
- [Derived] RENAL Replacement Therapy Study Investigators; Bellomo R, Cass A, Cole L, Finfer S, Gallagher M, Lo S, McArthur C, McGuinness S, Myburgh J, Norton R, Scheinkestel C, Su S. Intensity of continuous renal-replacement therapy in critically ill patients. N Engl J Med. 2009 Oct 22;361(17):1627-38. doi: 10.1056/NEJMoa0902413. PMID 19846848